CLINICAL TRIAL: NCT03341845
Title: Neoadjuvant AXITINIB and AVELUMAB for Patients With Localized Clear-cell RCC and a Moderate to High Risk
Brief Title: Neoadjuvant AXITINIB and AVELUMAB for Patients With Localized Clear-cell RCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N17JAV
Record Dates: First submitted 2017-11-09; First posted 2017-11-14 (Actual); Last update posted 2018-05-21 (Actual); Status verified 2018-04

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Axitinib; avelumab

STUDY DESIGN:
Intervention Model Description: simon's two stage design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- axitinib and avelumab (Experimental): axitinib 5MG BID and avelumab 10mg/kg Q2W
  Interventions: Drug: Axitinib; Drug: Avelumab

INTERVENTIONS:
Drug: Axitinib — axitinib in combination with avelumab
Drug: Avelumab — axitinib in combination with avelumab

SUMMARY:
a monocenter, open label, single arm, phase II study of the combination of axitinib with avelumab as neoadjuvant therapy in patients with intermediate to high-risk non-metastatic RCC.

DETAILED DESCRIPTION:
Renal cell carcinoma (RCC) accounts for 3% of adult malignancies and constitutes 95% of renal tumors. Surgical complete resection is currently the only curative treatment of RCC, including patients with locally advanced RCC or limited metastatic disease. However, these patients carry a high risk to develop locally recurrent disease and systemic progression. High risk patients with no evidence of disease following complete resection may therefore benefit from adjuvant and neo-adjuvant systemic treatment strategies which primarily aim to prolong disease free (DFS) and ultimately overall survival (OS). Neoadjuvant studies are a unique opportunity to further investigate the way in which immune checkpoint inhibition works and to identify predictors of treatment response. Recent research on intratumoral immune components after pretreatment of human renal cell carcinoma suggest a potential synergism for TKI with anti-PD-L1 therapy that could be exploited. In terms of downsizing tumours by pretreatment, axitinib has been shown to be more effective than sunitinib when comparing trials that have been performed with each drug. However, the immunemodulatory effect of axitinib has been ill defined. Since axitinib and anti-PD-L1 therapy would make for a potential synergism, two phase Ib dose-finding studies to evaluate safety, pharmacokinetics and pharmacodynamics of avelumab, an anti-PD-L1 monoclonal antibody, or pembrolizumab, an anti-PD1 monoclonal antibody, in combination with axitinib were performed. First results on response rate and safety profile presented at ESMO 2016 were promising with objective response rates of 67-70 % and toxicity profiles as seen with VEGFR-treatment. The investigator proposes a monocenter, open label, single arm, phase II study of the combination of axitinib with avelumab as neoadjuvant therapy in patients with intermediate to high-risk non-metastatic RCC. The statistical calculation of the primary endpoint is based on efficacy on the local tumour. The safety of this combination prior to surgery will be an important secondary endpoint.

ELIGIBILITY:
Inclusion Criteria:

Signed and written informed consent

* Male or female patients age ≥ 18 years
* Histologically confirmed diagnosis of non-metastatic clear-cell renal cell carcinoma of intermediate to high risk with completely resectable primary tumours.
* World Health Organization performance status of 0-1.
* Adequate coagulation function as defined in protocol
* Adequate hematological function as defined in protocol
* Adequate hepatic function as defined in protocol
* Adequate renal function as defined in protocol
* Negative serum pregnancy test at screening for women of childbearing potential.
* Highly effective contraception for both male and female subjects if the risk of conception exists.

Exclusion Criteria:

Renal tumors of low risk or M1

* Non-clear cell histology at biopsy
* Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product
* Corrected QT interval (QTc) > 480 msecs
* History of any of the cardiovascular conditions defined in the protocol within the past 6 months
* Poorly controlled hypertension
* History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months.
* Major surgery or trauma within 28 days prior to first dose of investigational product and/or presence of any non-healing wound, fracture, or ulcer
* Evidence of active bleeding or bleeding diathesis.
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures.
* Unable or unwilling to discontinue use of prohibited medications to be listed in protocol for at least 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of study drug and for the duration of the study
* Treatment with any of the following anti-cancer therapies: chemotherapy, immunotherapy, biologic therapy, investigational therapy or hormonal therapy within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of axitinib or avelumab
* Administration of any non-oncologic investigational drug within 30 days or 5 half lives whichever is longer prior to receiving the first dose of study treatment
* Prior organ transplantation, including allogeneic stem cell transplantation
* Significant acute or chronic infections as defined in protocol
* Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent
* Known severe hypersensitivity reactions to monoclonal antibodies
* Pregnancy or lactation
* Known alcohol or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-03-28 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
number of patients with partial remission | week 12 of neoadjuvant treatment
  according to RECIST 1.1.

SECONDARY OUTCOMES:
toxicity | up to 90 days after end of treatment
  measured by number and grade of adverse events
event free survival and overall survival | assessed up to 10 years
  Time from registration to disease progression or death

CONTACTS AND LOCATIONS:
Overall Officials: Axel Bex, MD, Principal Investigator — NKI-AvL
Locations (1):
- Antoni van Leeuwenhoek, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
decided by PI at each request for data

REFERENCES:
- [Derived] Bex A, van Thienen JV, Schrier M, Graafland N, Kuusk T, Hendricksen K, Lagerveld B, Zondervan P, van Moorselaar JA, Blank C, Wilgenhof S, Haanen J. A Phase II, single-arm trial of neoadjuvant axitinib plus avelumab in patients with localized renal cell carcinoma who are at high risk of relapse after nephrectomy (NEOAVAX). Future Oncol. 2019 Jul;15(19):2203-2209. doi: 10.2217/fon-2019-0111. Epub 2019 Apr 26. PMID 31023100